CLINICAL TRIAL: NCT03131856
Title: A Multidisciplinary Nutritional Intervention Programme Across Sectors to Improve the Nutritional Status of Geriatric Patients at Nutritional Risk - A Randomized Controlled Trial.
Brief Title: Nutritional Intervention in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Terp, Principal Investigater, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Geriatric-Project-2012
Record Dates: First submitted 2017-03-31; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Malnutrition
Keywords: Geriatrics; Nutritional risk; Multi-disciplinary intervention; Randomized Controlled Trial
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Eligible patients were randomized to either the intervention group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional intervention programme (Experimental): An individual dietary plan conducted by a clinical dietician before discharge in combination with three follow-up visits after discharge (1, 4 and 8 weeks).
  Interventions: Behavioral: Nutritional intervention programme
- Usual care (No Intervention): Usual care which means no individual dietary plan and no nutrition follow-up visits after discharge.

INTERVENTIONS:
Behavioral: Nutritional intervention programme — The intervention consisted of an individual dietary plan conducted by a clinical dietician before discharge in combination with three follow-up visits after discharge (1, 4 and 8 weeks) conducted by a district nurse.
  Arms: Nutritional intervention programme

SUMMARY:
This study aims to investigate the effect of a multi-disciplinary nutritional intervention program in geriatric nutritional at risk patients. The study is carried out as randomized controlled trial. The intervention consists of an individual dietary plan conducted by a clinical dietician before discharge in combination with three follow-up visits after discharge (1, 4 and 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or above
* BMI <20.5 and/or weight loss within the last 3 months and/or a reduced dietary intake in the previous week and/or severely ill

Exclusion Criteria:

* Terminal illness
* Active cancer diagnosis
* Permanently living in a nursing home
* Not willing or able to give an informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2015-08-17 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Three months follow-up
  Change in body weight (kg)

SECONDARY OUTCOMES:
Functional status | Three months follow-up
  Barthel Index (scale 0-100)
Functional status | Three months follow-up
  Handgrip strength (kg)
Self-rated health | Three months follow-up
  Self-rated health was measured with one single question with 5 possible responses on a Likert scale: In general, how would you rate your Health?
Re-admission | Up to three months
  All-cause unplanned readmissions
Mortality | 1) Up to 90 days after discharge 2) Up to 120 days after discharge
  All-cause mortality

IPD SHARING:
Plan to Share IPD: No